CLINICAL TRIAL: NCT04810390
Title: Multi-centre, Randomised, Double Blind, Placebo-controlled, Parallel, Phase III Study to Assess the Safety, Tolerability and Efficacy of Bilastine Ophthalmic Solution 0.6% in Children
Brief Title: Study to Assess the Safety, Tolerability and Efficacy of Bilastine Ophthalmic Solution 0.6% in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Collaborators: Dynamic Science S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BOFT-0520/PED
Record Dates: First submitted 2021-03-01; First posted 2021-03-23 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2022-07

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — bilastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilastine (Experimental): Daily instillation of one drop in each eye of Bilastine ophthalmic solution 0.6% for 8 weeks.
  Interventions: Drug: Bilastine
- Placebo (Placebo Comparator): Daily instillation of one drop in each eye of placebo for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bilastine — Ophthalmic solution 0.6%
  Arms: Bilastine
Drug: Placebo — Ophthalmic solution
  Arms: Placebo

SUMMARY:
This is a multi-centre, randomised, double blind, placebo-controlled, parallel-group, phase III study to assess the safety, tolerability and efficacy of Bilastine ophthalmic solution 0.6% in children with a documented history of seasonal allergic conjunctivitis (SAC) or perennial allergic conjunctivitis (PAC).

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients from 2 to under 18 years of age at V1a.
* 2. Documented history of AC before V1a.
* 3. Documented positive skin prick test and/or positive validated IgE test to seasonal (e.g. grass, ragweed, and/ or tree pollen) and/or perennial allergen (e.g. cat dander, dog dander, dust mites and/ or cockroach) within 6 months before V1a or a positive skin prick test at V1a.
* 4. Signs and symptoms of AC, i.e. tearing, itching and redness, that are likely to continue for the next weeks. Minimum score of four (in at least one eye) on an 11-item numeric rating scale in at least one of three categories at V1a.
* 5. Understanding of functioning and willingness to use e-diary at V1b and throughout study duration.
* 6. Willing to comply in all aspects of the study, including:

  1. use of IMP from V1b to V5a
  2. attending scheduled visits and completing telephone interviews.
* 7. Signed age-appropriate assent form (in participants 12 years of age and older) and written informed consent by the LAR in all cases. If a patient turns 18 years old during the clinical trial, a new written informed consent form will be provided and signed by the patient if he/she is willing to continue participating in the study.
* 8. Be able to self-administer eye drops satisfactorily or have a caregiver or LAR routinely available for this purpose. If a caregiver or LAR will be in charge of administering eye drops then he/she must attend Visit 1b, in order to be trained for administration of eye drops on-site.
* 9. For females of childbearing potential only: willingness to perform pregnancy tests, acceptance to use highly effective methods of birth control throughout the study duration. Highly effective methods of birth control include: combined hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner (provided that partner is the sole sexual partner of the clinical trial participant and has documentation of azoospermia) or sexual abstinence (if defined as refraining from heterosexual intercourse during the entire period of risk associated with the clinical trial treatment). The investigator is responsible for determining whether the subject has adequate birth control for study participation.

Exclusion Criteria:

* 1. History of known contraindications or sensitivities to the use of the IMPs or any of their components.
* 2. History of intraocular surgery within the previous 2 years before V1a, or planned surgery during study participation and within 2 weeks after follow-up.
* 3. History of ocular trauma (within the previous 6 months before V1a).
* 4. History or clinical evidence of ocular herpes simplex or ocular herpes zoster infectious disease within the previous year before V1a.
* 5. History of any clinically significant external ocular disease within 30 days before V1a.
* 6. Presence of dry eye, active blepharitis, active Meibomian gland dysfunction, active rosacea affecting the ocular surface/ lid margin, active or chronic follicular conjunctivitis, preauricular adenopathy, or any other ocular or periocular abnormality that may affect study outcome at V1a.
* 7. Known history of recurrent corneal erosion syndrome (idiopathic or secondary to dry eye).
* 8. History of treatment failure to topical antihistamines.
* 9. Prior (within 2 years before V1a), current or anticipated anti-allergy immunotherapy.
* 10. Prior (within 4 weeks before V1a), current or anticipated corticosteroid treatment (systemic or local, in case of depot-corticosteroids: within 6 weeks before V1a).
* 11. Prior (within 1 week before V1a), current or anticipated use of any ophthalmic agents (including artificial tears), except IMPs (starting at V1b).
* 12. Wearing of contact lenses 24 hours before ophthalmologic tests (V1a) and during clinical trial participation until V6.
* 13. Prior (within 2 weeks before V1a), current or anticipated systemic or intranasal treatment for allergic rhinitis.
* 14. Persons committed to an institution by virtue of an order issued either by the judicial or other authorities.
* 15. Pregnant woman, breastfeeding woman or woman planning a pregnancy.
* 16. Body weight below the 5th percentile for their age (patients 10 years of age or younger only).
* 17. Patient has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 30 days before V1a or is currently enrolled in an investigational interventional study.
* 18. Any condition that, in the opinion of the investigator, may jeopardise the clinical trial conduct according to the protocol. (For example, evidence of diseases, medications or laboratory abnormalities that could alter the conduct of the study).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of related ocular treatment-emergent adverse events (ocular r-TEAEs) | 8 weeks
  It will be reported the incidence of related ocular treatment-emergent adverse events (ocular r-TEAEs) as primary safety endpoint.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | 8 weeks
  It will be reported the incidence of treatment-emergent adverse events (TEAEs)
Incidence of ocular treatment-emergent adverse events (ocular TEAEs) | 8 weeks
  It will be reported the incidence of ocular treatment-emergent adverse events (ocular TEAEs)
Incidence of related treatment-emergent adverse events (r-TEAEs) | 8 weeks
  It will be reported the incidence of related treatment-emergent adverse events (r-TEAEs)
Incidence of abnormal clinical findings from ophthalmic examinations after instillation of IMP | 8 weeks
  It will be reported the incidence of abnormal clinical findings from ophthalmic examinations after instillation of IMP.
  Ophthalmic examination will consist of:
  * Best-corrected visual acuity test with age-appropriate techniques
  * Slit lamp biomicroscopy
  * Intraocular pressure in children who can cooperate with the test and do not require general anaesthesia
  * Non-dilated fundus examination
Mean peak ocular discomfort score after on-site instillation of IMP | 8 weeks
  Potential peak ocular discomfort caused by IMPs will be evaluated separately for each eye by the patient, with the aid of LAR if required, immediately upon instillation, on an 11-item numeric rating scale (from 0 to 10), which will include age-appropriate visual scales for children.
Mean ocular burning, stinging, tearing, blurring and stickiness scores after on-site instillation of IMP | 8 weeks
  Ocular tolerability (burning, stinging, tearing, blurring, and stickiness) of IMPs will be assessed separately for each eye by the patient with the aid of LAR if required,on an 11-item numeric rating scale (from 0 to 10), which will include age-appropriate visual scales for children.
Absolute value as well as absolute and relative changes from baseline of average daily total eye symptoms score (TESS) over the entire 8-week treatment period | 8 weeks
  The total eye symptoms score (TESS) based on the patient's e-diary is defined as the sum of the ocular itching, redness, and tearing scores. For each patient the worst daily sum of ratings will be selected for analysis. Additional exploratory analyses will be performed for each ocular symptom using the mean results of both eyes.
Absolute value as well as absolute and relative changes from baseline of average daily TESS at each week of the 8-week treatment period | 8 weeks
  The total eye symptoms score (TESS) based on the patient's e-diary is defined as the sum of the ocular itching, redness, and tearing scores. For each patient the worst daily sum of ratings will be selected for analysis. Additional exploratory analyses will be performed for each ocular symptom using the mean results of both eyes.
Absolute value as well as absolute and relative changes from baseline of average daily itching, redness and tearing scores over the entire 8-week treatment period | 8 weeks
  The average value for both eyes in each single symptom score will be used.
Absolute value as well as absolute and relative changes from baseline of average daily itching, redness and tearing scores at each week of the 8-week treatment period | 8 weeks
  The average value for both eyes in each single symptom score will be used.
For seasonal allergic conjunctivitis (SAC) patients only, the average daily TESS over the 2-week period of peak total eye symptoms score | 8 weeks
  For SAC patients, the average daily TESS and single symptom scores over the 2-week period of peak TESS and the 2-week period of peak single symptom scores, respectively, will be analysed using ANOVA.
For seasonal allergic conjunctivitis (SAC) patients only, the average daily itching, redness and tearing scores over the 2-week period of peak symptoms score | 8 weeks
  For SAC patients,the average daily itching, redness and tearing scores over the 2-week period of peak symptoms scores, respectively, will be analysed using ANOVA.

CONTACTS AND LOCATIONS:
Locations (18):
- Spain (18):
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Instituto Oftálmologico Quironsalud A Coruña, A Coruña
  - Hospital Universitari German Trias i Pujol (HGTiP),, Badalona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital General La Mancha Centro, Ciudad Real
  - Clínica Universidad de Navarra (CUN)- Sede Madrid, Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid
  - Hospital Quirónsalud Marbella, Marbella
  - Hospital Quirónsalud Málaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Clínica Juaneda, Palma de Mallorca
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario Donostia, San Sebastián
  - Hospital de Dia Quirónsalud Ave María, Seville
  - Hospital Quirón Valencia, Valencia
  - Hospital Universitario Dr. Peset Aleixandre, Valencia
  - Hospital Universitario Araba, Vitoria-Gasteiz